CLINICAL TRIAL: NCT06322303
Title: Effect of Cannabidiol (CBD) Consumption on Visual Function and Driving Performance
Brief Title: Effect of Cannabidiol (CBD) on Vision and Driving
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Sonia Ortiz Peregrina, Assistant Professor, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: C-EXP-194-UGR23
Record Dates: First submitted 2024-02-29; First posted 2024-03-21 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Cannabis Use
Keywords: cannabis; cannabidiol; vision; driving performance
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (CBD 0%) (Placebo Comparator): Participants are required to vaporize a placebo at 0% CBD concentration
  Interventions: Other: Placebo (CBD 0%)
- CBD 15% (Experimental): Participants are required to vaporize CBD at a concentration of 15%.
  Interventions: Other: CBD 15%
- CBD 30% (Experimental): Participants are required to vaporize CBD at a concentration of 30%.
  Interventions: Other: CBD 30%

INTERVENTIONS:
Other: Placebo (CBD 0%) — Participants are required to vaporize placebo at 0% CBD concentration
  Arms: Placebo (CBD 0%)
Other: CBD 15% — Participants are required to vaporize CBD at a concentration of 15%.
  Arms: CBD 15%
Other: CBD 30% — Participants are required to vaporize CBD at a concentration of 30%.
  Arms: CBD 30%

SUMMARY:
The use of cannabis with ∆9-tetrahydrocannabinol (THC) content has been shown to have negative effects on vision and driving. The use of other cannabinoids, such as cannabidiol (CBD), which is not attributed with a psychoactive effect, is increasing significantly. This project aims to investigate whether consuming CBD can negatively affect visual function by assessing a wide range of visual parameters and whether these changes may pose a risk for everyday activities such as driving.

ELIGIBILITY:
Inclusion Criteria:

* Being an occasional cannabis and/or cannabidiol user
* Have a current driving licence
* Have at least one year's driving experience
* Drive at least once a week
* Monocular visual acuity of at least 6/6 (Snellen) with habitual correction for driving
* Absence of binocular disorders

Exclusion criteria:

* Certain past or present medical conditions
* Current cannabis or alcohol use disorder
* Use of other drugs
* Pregnancy or lactation
* Simulator sickness.

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Overall Driving Performance Score (ODPS) after cannabidiol vaporization | Participants are assessed 20 minutes after vaporization
  To obtain the ODPS, Z-scores were calculated from individual parameters such as the standard deviation of the lateral lane position or the distance travelled into the opposite lane. The z-score is defined as a measure of how many standard deviations an individual value is below or above the group mean. The average Z-score of the individual driving variables is called the ODPS.
Change in motion detection sensitivity after cannabidiol vaporization | Participants are assessed 20 minutes after vaporization
  The subject has to indicate the direction of movement of a pattern of moving dots. The percentage of correct answers is obtained for different degrees of coherence.
Change in contrast sensitivity after cannabidiol vaporization | Participants are assessed 20 minutes after vaporization
  Contrast thresholds are obtained for different spatial frequencies
Change in visual acuity after cannabidiol vaporization | Participants are assessed 20 minutes after vaporization
  Visual acuity is assessed with a commercial test for distance vision.
Change in fixations after cannabidiol vaporization | Participants are assessed 20 minutes after vaporization
  The number of fixations made on different stimuli of interest in a task environment is counted using an eye tracker system.

SECONDARY OUTCOMES:
Driving simulator: standard deviation of the lateral lane position (SDLP) | Participants are assessed 20 minutes after vaporization
Distance travelled outside the lane | Participants are assessed 20 minutes after vaporization
  The SDLP assesses the lane weaving that the subject performs in the lane and indicates whether the vehicle's position is consistent.
Mean speed | Participants are assessed 20 minutes after vaporization
  Average speed is obtained and analyzed in relation to the speed limits for different sections.
Angular velocity of the steering wheel | Participants are assessed 20 minutes after vaporization
  The angular velocity of the steering wheel is a metric that indicates the subject's ability to maintain the vehicle's position.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Granada, Granada, Spain